CLINICAL TRIAL: NCT02173106
Title: Opportunity, Validity and Security of Steroids Plus Cyclosporin Therapy for Patients of Idiopathic Membranous Nephropathy : A Prospective, Randomized, Controlled, Multi-Center Clinical Trial
Brief Title: A Controlled Study of Steroids Plus Cyclosporin Therapy for Patients of Idiopathic Membranous Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, The Sixth Affiliated Hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usix-IMN-001
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Idiopathic Membranous Nephropathy; Proteinuria; Spontaneous Remission; Steroid Nephropathy; Cyclosporin Overdose
MeSH Terms: conditions — Glomerulonephritis, Membranous; Proteinuria; Remission, Spontaneous | interventions — Steroids; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A: steroid & Cyclosporin (Experimental): oral methylprednisolone 0.4mg/kg/d and 3.5~5mg/kg/d cyclosporin for 6 months.
  Interventions: Drug: steroid & Cyclosporin
- Group B: no steroid & Cyclosporin (No Intervention): no steroid and cyclosporin and waiting for spontaneous remission for 6 months

INTERVENTIONS:
Drug: steroid & Cyclosporin — oral methylprednisolone 0.4mg/kg/d and Cyclosporin for 6 months
  Arms: Group A: steroid & Cyclosporin

SUMMARY:
This prospective, randomized, controlled, multicenter clinical trial will evaluate Opportunity, Validity and Security of Steroids Plus Cyclosporin therapy for patients of Idiopathic Membranous Nephropathy.

DETAILED DESCRIPTION:
Idiopathic membranous nephropathy is a main reason for nephropathy. Since it can get spontaneous remission, in KDIGO, it is recommend that initial therapy should be started only in patients with nephrotic syndrome and when at least the following condition is met:urinary protein excretion persistently exceeds 4g/d and remains at over 50% of the baseline value,and does not show progressive and antiproteinuric therapy during an observation period of at least 6 months. But many retrospective researches reported that using steroids and immunosuppressive agents were better than waiting for spontaneous remission. There were few prospective, randomized, controlled research on whether it is better that begin to use steroids and immunosuppressive agent early without waiting for 6 months. In our study,we evaluate the validity and security of steroids plus cyclosporin therapy in idiopathic membranous nephropathy. This will be a prospective, randomized, controlled, multicenter study. Patients in treatment group will receive oral methylprednisolone 0.4mg/kg/d and 3.5~5mg/kg/d cyclosporin for 6 months. Patients in control group will waiting for spontaneous remission for 6 months,if there were no spontaneous remissions, patients in control group will receive oral methylprednisolone 0.4mg/kg/d and 3.5~5mg/kg/d cyclosporin for 6 months. After followed-up for 6 months the curative and side effect of steroid plus cyclosporin therapy in the early stage of idiopathic membranous nephropathy will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 14~75 years, regardless of gender without secondary reason, idiopathic membranous nephropathy by renal biopsy
* Average urinary protein excretion of at least3.5g/24h on two successive examinations,or plasma albumin <30g/l
* eGFR≥40ml/min/1.73m2
* Willingness to sign an informed consent

Exclusion Criteria:

* Secondary membranous nephropathy such as systemic lupus erythematosus, hepatitis B -associated nephritis
* Current or recent (within 30 days) exposure to high-dose of steroids or immunosuppressive therapy (CTX、MMF、CsA、FK506).
* Cirrhosis, chronic active liver disease
* History of significant gastrointestinal disorders (e.g. severe chronic diarrhea or active peptic ulcer disease)
* Any Active systemic infection or history of serious infection within one month.
* Other major organ system disease (e.g. serious cardiovascular diseases including congestive heart failure, chronic obstructive pulmonary disease, asthma requiring oral steroid treatment or central nervous system diseases)
* Active tuberculosis
* Known allergy, contraindication or intolerance to the steroids
* Pregnancy or breast feeding at the time of entry or unwillingness to comply with measures for contraception
* Malignant tumors
* Excessive drinking or drug abuse
* Mental aberrations
* Current or recent (within 30 days) exposure to any other investigational drugs

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Remission of proteinuria (complete or partial) | up to 6 months

SECONDARY OUTCOMES:
Deterioration of renal function (evidenced by a 50% rise from baseline serum creatinine (SCr) levels, or a 25% decline from baseline eGFR levels, or onset of end-stage renal disease or dialysis treatment, or kidney transplantation). | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zongpei Jiang, MD &Ph.D, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (6):
- China (6):
  - Department of Nephrology,Dongguan People's Hospital, Dongguan, Guangdong
  - Department of Nephrology, 2nd Affiliated Hospital,Guangzhou Medical University, Guangzhou, Guangdong
  - Department of Nephrology, 6th Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Department of Nephrology,Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - Department of Nephrology,1st Affiliated Hospital,Shenzhen University, Shenzhen, Guangdong
  - Department of Nephrology,1st People's Hospital of Zhaoqing, Zhaoqing, Guangdong

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952